CLINICAL TRIAL: NCT00538382
Title: Phase I Study of Pharmacokinetics and Pharmacodynamics of Artesunate in Pregnant Women in the Democratic Republic of Congo
Brief Title: Study of Pharmacokinetics and Pharmacodynamics of Artesunate in Pregnant Women in the Democratic Republic of Congo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of North Carolina (Other); Kinshasa School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: GN02- PK/PD of artesunate
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Malaria
Keywords: Malaria; Pregnancy; Artesunate; Pharmacokinetics; Pharmacodynamics; Democratic Republic of Congo
MeSH Terms: conditions — Malaria | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Case (Experimental): Cases are defined as parasitemic pregnant women during the second trimester (22-26 weeks gestation) and the third trimester (32-36 weeks gestation).
  Interventions: Drug: Artesunate
- Non-pregnant Control (Active Comparator): Non-pregnant controls are defined as parasitemic non-pregnant women recruited from the same community as the cases.
  Interventions: Drug: Artesunate
- Internal Control (Active Comparator): Internal controls are defined as the same women(cases)at three months postpartum.
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — A 200 mg dose of orally administered artesunate at the beginning of a 48-hour clinical sampling period.
  Other Names: Arsumax®

SUMMARY:
The objective of this study is to assess the pharmacokinetics (PK) and pharmacodynamics (PD) of a standard dose of orally administered artesunate, in order to determine if the current adult dose (200 mg) is appropriate in parasitemic pregnant women when compared to the same women at three months postpartum and to parasitemic non-pregnant women. Preliminary evidence on safety, tolerability and efficacy will be gathered.

DETAILED DESCRIPTION:
Annually, approximately 25 million African women become pregnant and are at risk of Plasmodium falciparum malaria infection during pregnancy [WHO]. The adverse effects of malaria during pregnancy include increased risk of maternal anemia, low birth weight (LBW) and infant death. The World Health Organization (WHO) recommends that intermittent preventive treatment (IPT) of malaria be used routinely in pregnant women living in areas of Africa where malaria infection is endemic. IPT involves the periodic presumptive administration of antimalarial treatment to all pregnant women as part of routine antenatal care.

This strategy has proven to be effective in much of sub-Saharan Africa where diagnostic facilities are often unavailable and pregnant woman are at high risk for malaria infection [WHO 2005]. This is representative of our study site in Kinshasa, Democratic Republic of Congo (DRC), where a 2004 pilot study conducted by the Global Network for Women's and Children's Health Research (GN) revealed that the prevalence of malaria in pregnant women was 34.3% [personal communication, Tshefu]. Currently sulfadoxine-pyrimethamine (SP) is the WHO-recommended drug for prevention of malaria during pregnancy where transmission of Plasmodium falciparum malaria is stable and where resistance to SP is low.

The DRC is an area of stable malaria transmission. In stable areas of transmission, non-pregnant adults have high levels of immunity to malaria and usually do not become severely ill with infection. However, pregnant women, especially primigravidas, have increased susceptibility to malaria. Pregnant women are not protected by immunity acquired in the non-pregnant state because parasites are exposed to different antigens in pregnancy than in the non-pregnant state. In addition, Plasmodium falciparum infection in pregnancy can lead to anemia and can affect placental nutrient transport, resulting in the birth of low birth weight infants with an increased risk for infant mortality [Steketee, 2001]. In a 2004 pilot study conducted by the Global Network in two large maternity clinics in Kinshasa, DRC, 34.3% (182/530) of pregnant women were thick smear positive for malaria [personal communication, Tshefu].

Currently, in Kinshasa, DRC the standard of care for IPT treatment of malaria during pregnancy is to administer 1500 mg sulfadoxine with 75 mg pyrimethamine during the second trimester (after the fourth month and usually in association with the mother's report of fetal quickening) and again during the third trimester, between 28-32 weeks gestation. SP has proven to be safe when used as IPT in pregnant women; clinical studies have shown no serious adverse events or cases of kernicterus nor has there been a significant difference in the rate of spontaneous abortions, premature deliveries, or neonatal deaths between IPT/SP and other interventions [Newman, 2004].

Since the 1980's, SP resistance in Africa and Asia has been steadily increasing. The 1999-2000 data from the East African Network for Monitoring Anti-malarial Treatment indicated that in vivo SP failure at some sites in Kenya was greater than 25% and had reached 45% at one site in Tanzania. Focal areas of low- to moderate-level SP resistance exist throughout Africa [Bilj, 2000; Deloron 1989; Landgraf, 1994; Nizla, 2000]. Resistance is likely to progress geographically and rapidly if nothing is done to interrupt this course. One of the reasons for the increasingly high SP failure rates may be the recently observed cross-resistance between SP and cotrimoxazole (sulfamethoxazole-trimethoprim) in Plasmodium falciparum [Lyer, 2001]. A second possible reason is that the long half-life of the drug may result in prolonged maintenance of subtherapeutic concentrations of the drug in the plasma [Nzila, 2000].

Resistance of Plasmodium falciparum to SP in Kinshasa appears to be low, but on the verge of increasing with selective pressure. In 2000, an in vivo drug efficacy trial in children found that 94.5% of the subjects responded adequately to SP [Kazadi, 2003]. These results have been corroborated by the genotyping of clinical samples from pregnant women in the 2004 pilot study conducted by the Global Network in Kinshasa for molecular markers for drug resistance [personal communication, Tshefu]. Molecular markers are used to survey the development and evolution of drug resistance. SP resistance is associated with mutations in the genes DHFR and DHPS. Presence of a quintuplet mutation (51, 59, 108, 437, and 540) is most strongly associated with SP resistance. Only 4.1% of the clinical samples in the pilot study contained the quintuplet mutation, which suggests that drug resistance was minimal at the time the study was conducted. However, 33.2% of the samples were found to be one mutation away from having the quintuplet mutation, indicating that full SP resistance (5 mutations) is likely to occur soon. Therefore, if adequate selective pressure were applied, e.g. by widespread use of SP, as is currently being practiced in the DRC, the prevalence of the quintuplet mutation and treatment failure due to drug resistance would increase dramatically.

Drug resistance to SP has spread more rapidly in the eastern part of the DRC, some 2000 kilometers (km) from Kinshasa. A report from a 2001 in vivo drug efficacy study in Bukavu, located on the Rwandan border in Eastern DRC, reported that 85.0% of the children responded adequately to SP [Kazadi, 2003]; however, a subsequent drug efficacy study in Rutshuru, also located on the Rwanda/Uganda border of Eastern DRC approximately 200 km south of Bukavu, demonstrated that only 39.4% of children responded adequately to treatment [Kazadi, personal communication]. In addition, 43.4% of these clinical samples contained the quintuplet mutation [Alker, personal communication]. Given this rise in resistance to SP in eastern DRC and the likelihood of increased resistance in Kinshasa, it is necessary to begin to explore other alternatives for SP.

While the pharmacokinetics of artemisinin is well known in non-pregnant adults, little is known about the specific pharmacokinetics of artemisinin in pregnant women, particularly pregnant women in developing countries. Dosages of drugs often need to be adjusted because of physiological and metabolic changes associated with pregnancy. The aim of this study is to determine the most appropriate dosage of artesunate to use in pregnant women in order to begin to investigate artesunate and artesunate combinations as options for IPT.

ELIGIBILITY:
Inclusion Criteria for Cases:

* 2nd trimester (22-26 weeks) or 3rd trimester (32-36 weeks) of pregnancy, based on an ultrasound conducted at <22 weeks gestation (composite of BPD, HC, AC, FL)
* Singleton pregnancy documented by ultrasound
* Parasitemic (> 500 parasites/μl)
* Afebrile and asymptomatic
* Hematocrit ≥ 30%
* Negative HIV test result
* At least 18 years of age and less than 40 years of age
* Able to spend three days in the clinic following their laboratory screening visit and again at three months postpartum
* Willing to provide informed consent

Inclusion Criteria for Non-pregnant Controls:

* Negative urine pregnancy test
* Parasitemic (> 500 parasites/μl)
* Afebrile and asymptomatic
* Hematocrit ≥ 30%
* Negative Determine® HIV test result
* At least 18 years of age and less than 40 years of age
* Able to spend three days in the clinic following screening
* Willing to provide informed consent

Inclusion Criteria for Internal controls:

* Negative urine pregnancy test

Exclusion Criteria for Cases:

* Parasitemia > 300,000 parasites/μl or symptomatic malaria
* Medical contraindications to participation or medical disorders (known high blood pressure, diabetes, sickle cell disease or tuberculosis)
* Have taken artesunate or any medicine containing artesunate during the current pregnancy
* Have taken any antimalarial in the past two weeks
* Have taken any medication in the past two weeks other than antipyretics (e.g., acetyl- salicylic acid, acetaminophen), folic acid or iron
* Have a fetus with any ultrasonographically visible structural fetal abnormalities identified on entry by ultrasound
* Past or present pregnancy complications that would preclude participation in the study (gestational diabetes/diabetes, incompetent cervix, pre-eclampsia/ eclampsia, and high blood pressure)
* Between 32-36 weeks gestation and have already participated in the study at 22-26 weeks gestation

Exclusion Criteria for Non-pregnant Controls:

* Parasitemia > 300,000 parasites/μl or have symptomatic malaria
* Medical contraindications to participation or medical disorders (known high blood pressure, diabetes, sickle cell disease or tuberculosis)
* Have taken any antimalarial in the past two weeks
* Have taken any medication in the past two weeks other than antipyretics (e.g., acetyl- salicylic acid, acetaminophen), folic acid or iron

Exclusion Criteria for Internal Controls:

* Parasitemia > 300,000 parasites/μl or have symptomatic malaria
* Have taken antimalarial medication in the past two weeks.
* Have taken any medication in the past two weeks other than antipyretics (e.g., acetyl- salicylic acid, acetaminophen), folic acid or iron
* Pregnant

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Levels of the unbound active major metabolite, dihydroartemisinin (DHA), will be similar for parasitemic pregnant women during their 2nd and 3rd trimesters vs. the same women 3 months postpartum | 48 hours

SECONDARY OUTCOMES:
The levels of unbound DHA will be similar for parasitemic pregnant women (during the second and third trimesters) vs. parasitemic non-pregnant women. | 48 hours after drug administration
The pharmacokinetics of ARTS and total DHA will be similar for parasitemic pregnant women (during the second and third trimesters) vs. the same women three months postpartum and parasitemic non-pregnant women. | 48 hours after drug administration
The pharmacodynamics of therapy will be similar for parasitemic pregnant women (during the 2nd and 3rd trimesters) vs. parasitemic non-pregnant women. Pharmacodynamics will be determined by measuring the parasite clearance time (PCT), PC50, and PC90. | 48 hours after drug administration
The pharmacodynamics and pharmacokinetic outcomes (as elaborated above) will be similar between the 2nd and 3rd trimester in parasitemic pregnant women. | 48 hours after drug administration
Description of safety and tolerability of Artesunate in the target population (pregnant women in the 2nd and 3rd trimester). | 0ne year postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Carl Bose, M.D., Principal Investigator — University of North Carolina; Antoinette Tshefu, M.D., M.P.H., Principal Investigator — Kinshasa School of Public Health
Locations (1):
- Kingasani Maternity Clinic, Kinshasa, Democratic Republic of the Congo

REFERENCES:
- [Derived] Onyamboko MA, Meshnick SR, Fleckenstein L, Koch MA, Atibu J, Lokomba V, Douoguih M, Hemingway-Foday J, Wesche D, Ryder RW, Bose C, Wright LL, Tshefu AK, Capparelli EV. Pharmacokinetics and pharmacodynamics of artesunate and dihydroartemisinin following oral treatment in pregnant women with asymptomatic Plasmodium falciparum infections in Kinshasa DRC. Malar J. 2011 Feb 28;10:49. doi: 10.1186/1475-2875-10-49. PMID 21352601
- See also: Website of the Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: RTI International — http://www.rti.org